CLINICAL TRIAL: NCT04970927
Title: Investigation of the Effect of Covid-19 Pandemic on Children With Cerebral Palsy
Brief Title: The Effect of Pandemic on Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Sevda Adar (Other)
Responsible Party: Sponsor-Investigator, Sevda Adar, assistant professor, medical doctor, Afyonkarahisar Health Sciences University
Organization: Afyonkarahisar Health Sciences University (Other)
Other Study IDs: SASP21
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Palsy; Covid19
Keywords: Cerebral Palsy; Covid19; Pandemics
MeSH Terms: conditions — Cerebral Palsy; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral Palsy (CP), is the most common cause of physical disability that begins in childhood and lasts throughout life, affecting 1 in 500 newborns, with an estimated prevalence of 17 million worldwide.

Social isolation, economic conditions, interruption of treatments, etc. may cause physical, mental, behavioral and psychosocial changes in children with cerebral palsy. Discontinuing regular physiotherapy can worsen functional skills and cause complications in children with cerebral palsy. Our aim in this study is to investigate the sustainability of the treatments of children with cerebral palsy during the pandemic period, their physical and psychosocial effects, and the relationship between their parents' fear of covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children under the age of 18 with cerebral palsy who applied to our hospital between 01.01.2014-31.01.2021

Exclusion Criteria:

* Parents of Cerebral Palsy Patients over 18 years of age
* Parents who cannot be reached by phone
* Parents who do not agree to fill out the questionnaire

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Parents of children under the age of 18 with cerebral palsy who applied to our hospital between 01.01.2014-31.01.2021
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Evaluation Survey | First day
  A questionnaire form consisting of 19 questions and 3 parts prepared by the authors in the light of the information obtained during the clinical observation process of children with cerebral palsy will be used.

SECONDARY OUTCOMES:
Covid-19 Fear Scale | First day
  Parents' fear of COVID-19 will be evaluated with the COVID-19 fear scale consisting of 7 questions. The items of the scale were created on the basis of a comprehensive review of existing scales on fear, expert evaluations, and participant interviews.

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA ADAR, Principal Investigator — Afyonkarahisar Health Sciences University; PETEK ŞARLAK KONYA, Study Chair — Afyonkarahisar Health Sciences University; ALİ İZZET AKÇİN, Study Chair — Afyonkarahisar Health Sciences University
Locations (1):
- Sevda Adar, Merkez, Afyonkarahisar, Turkey (Türkiye)